CLINICAL TRIAL: NCT03067077
Title: A Prospective, Randomized Comparison of SMILE Surgery to Wavefront-guided LASIK Surgery
Brief Title: A Prospective, Contralateral, Eye to Eye Comparison of SMILE Surgery to LASIK Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Edward E. Manche, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39587
Record Dates: First submitted 2017-02-16; First posted 2017-03-01 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Myopia
Keywords: SMILE; LASIK; Myopia; Wavefront-guided
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SMILE (Active Comparator): SMILE surgery
  Interventions: Procedure: SMILE; Procedure: LASIK
- Wavefront-guided LASIK (Active Comparator): Wavefront-guided LASIK
  Interventions: Procedure: SMILE; Procedure: LASIK

INTERVENTIONS:
Procedure: SMILE — SMILE surgery
Procedure: LASIK — LASIK surgery

SUMMARY:
Subjects will undergo SMILE surgery in one eye and LASIK surgery in their other eye to correct myopia.

DETAILED DESCRIPTION:
Subjects will have a comprehensive eye examination once they express an interest in the study. This includes a slit lamp examination of the front of the eye and a dilated fundoscopic examination of the back of the eye. If there is any pathology noted that would exclude the subject from the study, then we will inform the patient and make an appropriate referral. if the subject is deemed appropriate for the study after a comprehensive examination included computerized videokeratography, then they can be enrolled. Subjects will undergo bilateral simultaneous eye surgery. Which eye is treated with the WFG-LASIK and which eye is treated with SMILE will be randomized so there is a 50% chance for either eye to receive one treatment. Subjects will be seen on the day of surgery, post op day one, one week, one month, three months, six months and one year. Subjects will receive topical antibiotics in each eye for one week following the procedure. Subjects will receive topical steroid ophthalmic drops for one week after treatment. Subjects will also receive topical antibiotic ophthalmic drops for four days after treatment. All of this is within the usual and customary standard of care for the treatment of subjects undergoing LASIK and SMILE surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 22 and older with healthy eyes. Nearsightedness between -0.75 diopters and -8.00 diopters.
* Subjects with up to 3.00 diopters of astigmatism.

Exclusion Criteria:

* Subjects under the age of 22.
* Subjects with excessively thin corneas.
* Subjects with topographic evidence of keratoconus.
* Subjects with ectatic eye disorders.
* Subjects with autoimmune diseases.
* Subjects who are pregnant or nursing.
* Subjects must have similar levels of nearsightedness in each eye. They can not be more than 1.5 diopter of difference between eyes.
* Subjects with 3.25 or more diopters of astigmatism
* Subjects must have similar levels of astigmatism in each eye. They can not have more than 0.50 diopters of difference between eyes.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-12 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Manche, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiang B, Valerio GS, Manche EE. Prospective, Randomized Contralateral Eye Comparison of Wavefront-Guided Laser In Situ Keratomileusis and Small Incision Lenticule Extraction Refractive Surgeries. Am J Ophthalmol. 2022 May;237:211-220. doi: 10.1016/j.ajo.2021.11.013. Epub 2021 Nov 14. PMID 34788593
- [Derived] Ma KK, Manche EE. Patient-reported quality of vision in a prospective randomized contralateral-eye trial comparing LASIK and small-incision lenticule extraction. J Cataract Refract Surg. 2023 Apr 1;49(4):348-353. doi: 10.1097/j.jcrs.0000000000001127. PMID 36539217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled participants were to receive SMILE surgery in one eye and LASIK surgery in their fellow eye
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | SMILE | Wavefront-guided LASIK
Started | 44; 44 Eyes | 44; 44 Eyes
Received Surgery | 40; 40 Eyes | 39; 39 Eyes
Completed | 37; 37 Eyes | 37; 37 Eyes
Not Completed | 7; 7 Eyes | 7; 7 Eyes
Not completed — Did not receive surgery | 4 | 5
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants receive SMILE surgery in one eye and Wavefront-guided LASIK in the fellow eye.
Arm/Group | All Participants
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 19
  Caucasian | 18
  Hispanic | 2
  Indian | 4
  Pacific Islander | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participant Eyes With an Uncorrected Visual Acuity of 20/20 or Better
Description: ETDRS testing lane
Time Frame: One year
Population: Participants who completed 12 month follow-up
Measure: Number; unit: percentage of participant eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
percentage of participant eyes | 94 | 83

2. Secondary Outcome: Number of Participant Eyes Losing 2 or More Lines of Corrected Distance Visual Acuity
Description: ETDRS testing lane
Time Frame: One year
Population: Participants who completed the 12 month follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes | 0 | 0

3. Secondary Outcome: Aberrometry Measurements
Description: Increase in total higher order RMS (root mean squared) by greater than 0.5 microns
Time Frame: One year
Population: Participants who completed 12 months follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes | 0 | 0

4. Secondary Outcome: Patient Satisfaction
Description: Percentage of patients satisfied with surgery. Patients were asked yes or no.
Time Frame: One year
Population: Participants who completed 12 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Participants | 36 | 36

5. Secondary Outcome: Change in Corneal Sensation
Description: A decrease in corneal sensation of more than 4 cm as measured by Cochet-Bonnet Aesthesiometry
Time Frame: One year
Population: Participants who completed 12 months follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes | 0 | 0

6. Secondary Outcome: Dry Eye Symptoms as Measured by OSDI Index
Description: Worsening of ocular surface disease index (OSDI) score of greater than 25. The overall OSDI score defined the ocular surface as normal (0-12 points) or as having mild (13-22 points), moderate (23-32 points), or severe (33-100 points) disease.
Time Frame: One year
Population: Patients who completed 12 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Participants | 0 | 0

7. Secondary Outcome: Analysis of Astigmatism
Description: Participant eyes with an increase in astigmatism of greater than 1.0 diopter
Time Frame: One year
Population: Participants with 12 months follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes | 0 | 0

8. Secondary Outcome: Anterior Segment Ocular Coherence Topography Analysis
Description: Humphrey Visante AS OCT
Time Frame: One year
Population: The outcome could not be analyzed because the data were corrupted
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Predictability
Description: Number of eyes within +/- 0.5 and +/- 1.00 diopter of the intended correction
Time Frame: One year
Population: Participants who completed 12 months follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes
  +/- 0.50 diopters | 30 | 34
  +/- 1.0 diopters | 36 | 37

10. Secondary Outcome: Stability
Description: Change in refractive error greater than one diopter over 1 to 12 months
Time Frame: One year
Population: Participants who completed twelve months follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | SMILE | Wavefront-guided LASIK
Number analyzed (Participants) | 37 | 37
Number analyzed (Eyes) | 37 | 37
Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events are reported per participant
Arm/Group | SMILE | Wavefront-guided LASIK
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 1/44 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMILE (N=44) | Wavefront-guided LASIK (N=44)
Unable to remove SMILE lenticule (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03067077/Prot_000.pdf